CLINICAL TRIAL: NCT05925153
Title: Vision Screening Study for College Students at Nankai University
Status: Completed | Type: Observational
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY2023030
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2022-09

CONDITIONS: Myoma
MeSH Terms: conditions — Myoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- College Students
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The prevalence of myopia among high school students in China is as high as 80%-90%. For college students with longer years of education, the majority of myopia and the factors influencing the prevalence of high myopia should be better understood for timely prevention and treatment. This study aims to investigate the prevalence of myopia and education-related influencing factors among college students at Nankai University.

ELIGIBILITY:
Inclusion Criteria:

* All 1st year students

Exclusion Criteria:

* No eye diseases such as cataracts, glaucoma,keratoconus, etc.
* No psychiatric disorders
* Astigmatism ≤ -6.00D

Ages: 16 Years to 30 Years | Sex: All
Age Groups: Child, Adult
Study Population: All 1st-year freshmen at Nankai University with no significant systemic or eye diseases are eligible for vision screening
Sampling Method: Non-Probability Sample
Enrollment: 8500 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of myopia | One day measurement
  Myopia was defined as an equivalent spherical refraction ≤ -0.50D in either eye
Prevalence of high myopia | One day measurement
  High myopia was defined as an equivalent spherical refraction ≤ -6.00D in either eye

SECONDARY OUTCOMES:
Blood pressure | One day measurement
  Venous blood pressure was measured using a sphygmomanometer, and systolic and diastolic blood pressure results were recorded.
Pulse | One day measurement
  Measure the number of pulses in the quiet state and record the number of beats per minute.

CONTACTS AND LOCATIONS:
Locations (1):
- Tiajin Eye Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wei S, Sun Y, Li S, Hu J, Yang X, Lin C, Cao K, Du J, Guo J, Li H, Wang N. Refractive Errors in University Students in Central China: The Anyang University Students Eye Study. Invest Ophthalmol Vis Sci. 2018 Sep 4;59(11):4691-4700. doi: 10.1167/iovs.18-24363. PMID 30267091
- [Background] Wei S, Sun Y, Li SM, Hu J, Cao K, Du J, An W, Liang X, Guo J, Li H, Wang N. Visual Impairment and Spectacle Use in University Students in Central China: The Anyang University Students Eye Study. Am J Ophthalmol. 2019 Oct;206:168-175. doi: 10.1016/j.ajo.2019.04.026. Epub 2019 May 10. PMID 31078530
- [Background] Huang L, Kawasaki H, Liu Y, Wang Z. The prevalence of myopia and the factors associated with it among university students in Nanjing: A cross-sectional study. Medicine (Baltimore). 2019 Mar;98(10):e14777. doi: 10.1097/MD.0000000000014777. PMID 30855486